CLINICAL TRIAL: NCT03688711
Title: A Randomized, Double-blind, Parallel-group Trial to Confirm the Clinical Efficacy and Safety of Dasiglucagon in the Rescue Treatment of Hypoglycemia in Subjects With Type 1 Diabetes Mellitus (T1DM) Compared to Placebo
Brief Title: Trial to Confirm the Clinical Efficacy and Safety of Dasiglucagon in the Treatment of Hypoglycemia in Subjects With T1DM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZP4207-17145
Record Dates: First submitted 2018-09-25; First posted 2018-09-28 (Actual); Results first posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Hypoglycemia; Diabetes Mellitus, Type 1
Keywords: glucagon
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1 | interventions — dasiglucagon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dasiglucagon (Experimental): single fixed dose (subcutaneous injection) of dasiglucagon
  Interventions: Drug: Dasiglucagon
- Placebo (Placebo Comparator): single fixed dose (subcutaneous injection) of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dasiglucagon — Glucagon analogue
  Other Names: ZP4207
  Arms: Dasiglucagon
Drug: Placebo — Placebo for dasiglucagon
  Other Names: Placebo for dasiglucagon
  Arms: Placebo

SUMMARY:
A randomized, double-blind, parallel-group trial to confirm the clinical efficacy and safety of dasiglucagon in the rescue treatment of hypoglycemia in subjects with type 1 diabetes mellitus (T1DM) compared to placebo

DETAILED DESCRIPTION:
Subjects were randomized in a ratio of 3:1 to receive a single subcutaneous dose of dasiglucagon (0.6 mg) or matching placebo. Randomization also determined whether the subject was to be injected in the buttock or deltoid. During the dosing visit (Visit 2), hypoglycemia was induced by a fast-acting insulin glulisine (Apidra®) infusion, and trial drug was administered when the subject's plasma glucose level was 45-60 mg/dL (2.5-3.3 mmol/L). During the insulin-induced hypoglycemia, pharmacokinetic and pharmacodynamic samples were drawn, and plasma glucose levels were monitored closely at site for safety reasons. A rescue glucose infusion could be administered to ameliorate persistent hypoglycemia. Subjects were followed for at least 28 days after dosing to perform an adequate immunogenicity evaluation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects with T1DM for at least 1 year; diagnostic criteria as defined by the American Diabetes Association (3).
* Treated with insulin for T1DM for at least 1 year and with stable insulin treatment (defined as no more than a 10-unit daily variation in total daily insulin dose) 30 days prior to screening
* Hemoglobin A1c <10%.
* Aged between 18 and 75 years, both inclusive.

Exclusion Criteria:

* Previous participation in a clinical trial within the dasiglucagon in the rescue treatment of hypoglycemia program.
* Known or suspected allergy to trial drug(s) or related products.
* History of anaphylaxis or symptoms of severe systemic allergy (such as angioedema).
* Previous participation in this trial. Participation being defined by signing the informed consent document.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Sylvest, MSc Pharm, Study Director — Zealand Pharma A/S
Locations (3):
- United States (3):
  - ProSciento, Inc., Chula Vista, California
  - AMCR Institute, Escondido, California
  - Rainier Clinical Research, Inc., Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasiglucagon 0.6 mg: single fixed dose (subcutaneous injection) of dasiglucagon
  Dasiglucagon: Glucagon analogue
Period: Overall Study
Arm/Group | Dasiglucagon 0.6 mg | Placebo
Started (Randomized) | 34 | 11
Completed | 34 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population of all randomized subjects who received at least one dose of trial drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasiglucagon 0.6 mg | Placebo | Total
Number analyzed (Participants) | 34 | 10 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (13.49) | 36.5 (12.80) | 41.0 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 1 | 19
  Male | 16 | 9 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 30 | 7 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 34 | 7 | 41
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 10 | 44
Body weight [Mean (Standard Deviation); unit: kg] | 84.49 (20.102) | 83.69 (10.812) | 84.30 (18.295)
Body mass index [Mean (Standard Deviation); unit: kg per square metre] | 28.41 (5.802) | 27.92 (3.975) | 28.30 (5.402)
Duration of diabetes [Mean (Standard Deviation); unit: years] | 22.5 (13.82) | 21.2 (13.42) | 22.2 (13.59)

OUTCOME MEASURES:

1. Primary Outcome: Time to Plasma Glucose Recovery.
Description: Plasma glucose recovery was defined as first increase in plasma glucose of ≥20 mg/dL (1.1 mmol/L) from baseline during the hypoglycemic clamp procedure without administration of rescue intravenous (IV) glucose. Patients who received rescue IV glucose before 45 minutes and patients not recovering within 45 minutes after dosing were censored at 45 minutes.
Time Frame: 0-45 minutes after dosing
Population: The full analysis set of all randomized subjects who received at least one dose of trial drug (same as the safety analysis set)
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Dasiglucagon 0.6 mg | Placebo
Number analyzed (Participants) | 34 | 10
minutes | 10.0 [8.0 to 12.0] | 35.0 [20.0 to NA] — The upper limit was not estimable due to insufficient number of participants reaching recovery
Statistical Analysis 1: Comparison: Dasiglucagon 0.6 mg vs Placebo; The recovery rates of dasiglucagon and placebo were evaluated using a Kaplan Meier (KM) approach, with treatment group as a stratification factor. Differences between the KM curves (dasiglucagon versus placebo) were evaluated inferentially using pairwise two-sided log-rank tests stratified by injection site; Test type: Superiority; p < 0.0001, Log Rank

2. Secondary Outcome: Plasma Glucose Recovery After Trial Drug Injection
Description: Plasma glucose recovery (patient has achieved increase in plasma glucose of ≥20 mg/dL (1.1 mmol/L)) within 30 minutes, within 20 minutes, within 15 minutes, and within 10 minutes after trial drug injection without administration of rescue intravenous (IV) glucose.
Time Frame: 0-30 minutes after dosing
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dasiglucagon 0.6 mg | Placebo
Number analyzed (Participants) | 34 | 10
Participants
  Glucose recovery within 30 minutes | 33 | 5
  Glucose recovery within 20 minutes | 32 | 1
  Glucose recovery within 15 minutes | 30 | 0
  Glucose recovery within 10 minutes | 21 | 0
Statistical Analysis 1: Comparison: Dasiglucagon 0.6 mg vs Placebo; Assessed at 30 minutes. The recovery rates of dasiglucagon and placebo were compared at each time point using a Fisher's exact test. Testing followed an a priori defined hierarchical inferential test order, proceeding until the first failure to reject the null hypothesis comparing dasiglucagon versus placebo; Test type: Superiority; p = 0.0012, Fisher Exact
Statistical Analysis 2: Comparison: Dasiglucagon 0.6 mg vs Placebo; Assessed at 20 minutes. The recovery rates of dasiglucagon and placebo were compared at each time point using a Fisher's exact test. Testing followed an a priori defined hierarchical inferential test order, proceeding until the first failure to reject the null hypothesis comparing dasiglucagon versus placebo; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 3: Comparison: Dasiglucagon 0.6 mg vs Placebo; Assessed at 15 minutes. The recovery rates of dasiglucagon and placebo were compared at each time point using a Fisher's exact test. Testing followed an a priori defined hierarchical inferential test order, proceeding until the first failure to reject the null hypothesis comparing dasiglucagon versus placebo; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 4: Comparison: Dasiglucagon 0.6 mg vs Placebo; Assessed at 10 minutes. The recovery rates of dasiglucagon and placebo were compared at each time point using a Fisher's exact test. Testing followed an a priori defined hierarchical inferential test order, proceeding until the first failure to reject the null hypothesis comparing dasiglucagon versus placebo; Test type: Superiority; p = 0.0006, Fisher Exact

3. Secondary Outcome: Plasma Glucose Changes From Baseline
Description: Plasma glucose changes from baseline at 30 minutes, at 20 minutes, at 15 minutes, and at 10 minutes after trial drug injection or at the time of rescue (patient level).
Time Frame: 0-30 minutes after dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dasiglucagon 0.6 mg | Placebo
Number analyzed (Participants) | 34 | 10
mg/dL
  At 30 minutes | 85.29 (29.696) | 15.14 (9.328)
  At 20 minutes | 52.95 (20.298) | 9.67 (8.846)
  At 15 minutes | 41.62 (17.077) | 5.23 (6.686)
  At 10 minutes | 24.54 (12.560) | 0.62 (6.100)
Statistical Analysis 1: Comparison: Dasiglucagon 0.6 mg vs Placebo; Change from baseline in plasma glucose at 30 minutes after investigational product injection was calculated using nominal sampling times and analyzed using an analysis of variance model with treatment, age group and injection site for each endpoint. Testing followed an a priori defined hierarchical inferential test order, proceeding until the first failure to reject the null hypothesis comparing dasiglucagon versus placebo; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Dasiglucagon 0.6 mg vs Placebo; Change from baseline in plasma glucose at 20 minutes after investigational product injection was calculated using nominal sampling times and analyzed using an analysis of variance model with treatment, age group and injection site for each endpoint. Testing followed an a priori defined hierarchical inferential test order, proceeding until the first failure to reject the null hypothesis comparing dasiglucagon versus placebo; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 3: Comparison: Dasiglucagon 0.6 mg vs Placebo; Change from baseline in plasma glucose at 15 minutes after investigational product injection was calculated using nominal sampling times and analyzed using an analysis of variance model with treatment, age group and injection site for each endpoint. Testing followed an a priori defined hierarchical inferential test order, proceeding until the first failure to reject the null hypothesis comparing dasiglucagon versus placebo; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 4: Comparison: Dasiglucagon 0.6 mg vs Placebo; Change from baseline in plasma glucose at 10 minutes after investigational product injection was calculated using nominal sampling times and analyzed using an analysis of variance model with treatment, age group and injection site for each endpoint. Testing followed an a priori defined hierarchical inferential test order, proceeding until the first failure to reject the null hypothesis comparing dasiglucagon versus placebo; Test type: Superiority; p < 0.0001, ANCOVA

4. Secondary Outcome: Time to Target Plasma Glucose Concentration
Description: Time to first plasma glucose concentration ≥70 mg/dL (3.9 mmol/L) without administration of rescue intravenous glucose
Time Frame: 0-45 minutes after dosing
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Dasiglucagon 0.6 mg | Placebo
Number analyzed (Participants) | 34 | 10
minutes | 9.0 [8.0 to 10.0] | 27.5 [12.0 to 40.0]
Statistical Analysis 1: Comparison: Dasiglucagon 0.6 mg vs Placebo; Evaluated using a Kaplan Meier (KM) approach, with treatment group as a stratification factor, analogous to that used for the primary endpoint analysis. Differences between the KM curves (dasiglucagon versus placebo) were evaluated inferentially using pairwise two-sided log-rank tests. Subjects whose time to first plasma glucose concentration ≥70 mg/dL (3.9 mmol/L) was not met within 45 minutes post-dosing were censored, at the time of the last valid plasma glucose measurement up to 45 minutes; Test type: Superiority; p < 0.0001, Log Rank

5. Secondary Outcome: Pharmacodynamics - Area Under the Effect Curve
Description: Plasma glucose response as area under the effect curve (AUE) above baseline from time zero to 30 minutes, AUE0-30min.
Time Frame: 0-30 minutes after dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*mg/dL
Arm/Group | Dasiglucagon 0.6 mg | Placebo
Number analyzed (Participants) | 34 | 10
hr*mg/dL | 19.9 (8.41) | 2.67 (3.06)
Statistical Analysis 1: Comparison: Dasiglucagon 0.6 mg vs Placebo; The analysis was an analysis of covariance (ANCOVA) model with treatment group as factor and the baseline of the dependent variable plasma glucose as a covariate; Test type: Superiority; p < 0.0001, ANCOVA; Odds Ratio (OR) = 4.05, 95% CI 2-sided [2.71 to 6.05]

6. Secondary Outcome: Pharmacokinetics - Area Under the Plasma Concentration Curve
Description: Area under the drug concentration curve (AUC) from time zero to 90 minutes, AUC0-90min
Time Frame: 0-90 minutes after dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pmol/L
Arm/Group | Dasiglucagon 0.6 mg
Number analyzed (Participants) | 34
hr*pmol/L | 1480 (34.6)

7. Secondary Outcome: Pharmacokinetics - Area Under the Plasma Concentration Curve
Description: Area under the drug concentration curve (AUC) from time zero to 120 minutes, AUC0-120min
Time Frame: 0-120 minutes after dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pmol/L
Arm/Group | Dasiglucagon 0.6 mg
Number analyzed (Participants) | 34
hr*pmol/L | 1780 (31.6)

8. Secondary Outcome: Pharmacokinetics - Maximum Plasma Concentration
Description: Maximum plasma dasiglucagon concentration (Cmax)
Time Frame: 0-120 minutes after dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | Dasiglucagon 0.6 mg
Number analyzed (Participants) | 34
pmol/L | 1350 (38.2)

9. Secondary Outcome: Pharmacokinetics - Time to Maximum Plasma Concentration
Description: Time to maximum plasma dasiglucagon concentration (tmax)
Time Frame: 0-120 minutes after dosing
Population: as for outcome 1
Measure: Median (Full Range); unit: minutes
Arm/Group | Dasiglucagon 0.6 mg
Number analyzed (Participants) | 34
minutes | 35 [15 to 60]

10. Secondary Outcome: Immunogenicity - Occurrence of Anti-drug Antibodies
Description: Occurrence of antibodies against dasiglucagon. Presented as percentage of patients with antibodies.
Time Frame: 58 days
Population: The safety analysis set of all randomized subjects who received at least one dose of trial drug (same as the full analysis set)
Measure: Count of Participants; unit: Participants
Arm/Group | Dasiglucagon 0.6 mg | Placebo
Number analyzed (Participants) | 34 | 10
Participants | 0 | 0

11. Secondary Outcome: Rescue Infusions of IV Glucose After Trial Drug Administration
Description: Presented as number of patients with rescue infusions of IV glucose after trial drug administration. This was a safety outcome measure. IV = intravenous
Time Frame: 0-45 minutes after dosing
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dasiglucagon 0.6 mg | Placebo
Number analyzed (Participants) | 34 | 10
Participants | 1 | 1

12. Secondary Outcome: Time to First Rescue Infusion of IV Glucose After Trial Drug Administration
Description: Safety outcome measure: time to first rescue infusion of IV glucose after trial drug administration. IV = intravenous
Time Frame: 0-45 minutes after dosing
Population: Only the patients who received IV glucose administration are included.
Measure: Number; unit: minutes
Arm/Group | Dasiglucagon 0.6 mg | Placebo
Number analyzed (Participants) | 1 | 1
minutes | 10 | 14

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Dasiglucagon 0.6 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/10
Other Adverse Events (participants affected / at risk) | 24/34 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasiglucagon 0.6 mg (N=34) | Placebo (N=10)
Nausea (Gastrointestinal disorders) | 21 (21) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (11) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 6 (29) | 2 (3)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 2 (2) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-04): https://cdn.clinicaltrials.gov/large-docs/11/NCT03688711/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT03688711/SAP_001.pdf